CLINICAL TRIAL: NCT05719428
Title: A Phase II Trial of Neural Network-based Treatment Decision Support Tool in Patients With Refractory Solid Organ Malignancies
Brief Title: Neural Network-based Treatment Decision Support Tool in Patients With Refractory Solid Organ Malignancies
Acronym: DRUID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: School of Computing, National University of Singapore (Unknown); National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/00653
Record Dates: First submitted 2023-01-30; First posted 2023-02-09 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Solid Organ Malignancies
Keywords: Next generation sequencing; DRUID

STUDY DESIGN:
Intervention Model Description: Patients NGS profile will be analysed with DRUID system to generate recommendations based on predicted efficacy. Patients with available archival tissue will have gene expression analysis performed to optimise DRUID recommendation. Patients will subsequently receive single agent therapy based on DRUID recommendations and criteria for therapy choice.
  Patients will begin single agent therapy within 4 weeks of enrolment and continue until disease progression, maximum safe cumulative dose reached (where applicable, per standard institution practice) or unacceptable toxicity as per physician's discretion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DRUID (Experimental): Patients NGS profile will be analysed with DRUID system to generate recommendations based on predicted efficacy. Patients with available archival tissue will have gene expression analysis performed to optimise DRUID recommendation. Patients will subsequently receive single agent therapy based on DRUID recommendations and criteria for therapy choice.
  Interventions: Other: DRUID AI Program

INTERVENTIONS:
Other: DRUID AI Program — Patients will begin single agent therapy within 4 weeks of enrolment and continue until disease progression, maximum safe cumulative dose reached (where applicable, per standard institution practice) or unacceptable toxicity as per physician's discretion.

SUMMARY:
DRUID is a treatment decision support tool combining predictive models and public databases related to multi-gene markers, drug response screens, gene essentiality and clinical status of drugs to provide drug recommendations personalized based on an input genomic profile. We hypothesize that DRUID analysis of patients' somatic mutational profile from NGS diagnostic platform can be used as a treatment decision support tool in patients with refractory cancer without targetable mutations.

DETAILED DESCRIPTION:
2.1. Hypothesis We hypothesize that DRUID analysis of patients' somatic mutational profile from NGS diagnostic platform can be used as a treatment decision support tool in patients with refractory cancer without targetable mutations. Using algorithm selected treatment from a panel of 60 drugs we predict an objective response rate (ORR) of ≥ 25%.

2.2. Primary Objectives

• To prospectively determine if DRUID selected therapy based on NGS diagnostic profile input can lead to objective responses in refractory solid organ malignancies.

2.3. Secondary Objectives

* To assess clinical benefit rate (complete response, partial response and stable disease for ≥ 24 weeks)
* To assess progression-free and overall survival of patients treated with DRUID-guided therapy

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet all of the following criteria:

* Age ≥ 21 years.
* Histological or cytological diagnosis solid organ malignancy
* Available results of comprehensive NGS panel testing performed on either tumour tissue or blood-based assay. If results are from blood-based assay, test must have been performed in the metastatic setting.
* ECOG 0-2.
* At least 1 measurable tumour lesions based on RECIST 1.1 criteria
* Estimated life expectancy of at least 12 weeks.
* Has documented progressive disease from last line of therapy.
* Has received at least 2 lines of palliative systemic therapy with no available standard therapy:
* Adequate organ function including the following:

  * Bone marrow:

    * Absolute neutrophil (segmented and bands) count (ANC) ≥ 1.5 x 109/L
    * Platelets ≥ 100 x 109/L
    * Haemoglobin ≥ 8 x 109/L
  * Hepatic:

    * Bilirubin ≤ 1.5 x upper limit of normal (ULN),
    * ALT or AST ≤ 2.5x ULN, (or ≤ 5 X with liver metastases)
  * Renal:

    * Creatinine ≤ 1.5x ULN
    * Signed informed consent from patient or legal representative.
* Able to comply with study-related procedures.

Exclusion Criteria:

* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumour therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Major surgery within 28 days of study drug administration.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Active bleeding disorder or bleeding site.
* Non-healing wound.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrolment.
* Symptomatic brain metastasis.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 10 months
  Defined as patient exhibiting a best study response of complete or partial clinical response based on radiological imaging per RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Clinical benefit | 10 months
  Defined as presence of best study response of complete or partial response or stable disease for at least 24 weeks (based on RECIST 1.1 criteria).
Progression free survival | From enrolment till disease progression or date of death or final follow-up visit (1 year).
  Defined as the time from the date of study enrolment to the first date of documented disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Robert John Walsh, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Department of Hematology-Oncology, National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hickcox JP. Treatment of fractures with Hirschhorn compression plates. J Am Vet Med Assoc. 1970 Jan 15;156(2):187-96. No abstract available. PMID 5461196
- [Background] Garraway LA, Verweij J, Ballman KV. Precision oncology: an overview. J Clin Oncol. 2013 May 20;31(15):1803-5. doi: 10.1200/JCO.2013.49.4799. Epub 2013 Apr 15. No abstract available. PMID 23589545
- [Background] Clerch AR, Miale JB. A comparison of the Unitest system with three other methods for determining blood glucose. Am J Clin Pathol. 1971 Feb;55(2):159-62. doi: 10.1093/ajcp/55.2.159. No abstract available. PMID 5541669
- [Background] Mariappan R, Jayagopal A, Sien HZ, Rajan V. Neural Collective Matrix Factorization for integrated analysis of heterogeneous biomedical data. Bioinformatics. 2022 Sep 30;38(19):4554-4561. doi: 10.1093/bioinformatics/btac543. PMID 35929808
- [Background] Nguyen T, Nguyen GTT, Nguyen T, Le DH. Graph Convolutional Networks for Drug Response Prediction. IEEE/ACM Trans Comput Biol Bioinform. 2022 Jan-Feb;19(1):146-154. doi: 10.1109/TCBB.2021.3060430. Epub 2022 Feb 3. PMID 33606633
- [Background] Garnett MJ, Edelman EJ, Heidorn SJ, Greenman CD, Dastur A, Lau KW, Greninger P, Thompson IR, Luo X, Soares J, Liu Q, Iorio F, Surdez D, Chen L, Milano RJ, Bignell GR, Tam AT, Davies H, Stevenson JA, Barthorpe S, Lutz SR, Kogera F, Lawrence K, McLaren-Douglas A, Mitropoulos X, Mironenko T, Thi H, Richardson L, Zhou W, Jewitt F, Zhang T, O'Brien P, Boisvert JL, Price S, Hur W, Yang W, Deng X, Butler A, Choi HG, Chang JW, Baselga J, Stamenkovic I, Engelman JA, Sharma SV, Delattre O, Saez-Rodriguez J, Gray NS, Settleman J, Futreal PA, Haber DA, Stratton MR, Ramaswamy S, McDermott U, Benes CH. Systematic identification of genomic markers of drug sensitivity in cancer cells. Nature. 2012 Mar 28;483(7391):570-5. doi: 10.1038/nature11005. PMID 22460902
- [Background] De Lange T, Kooter JM, Michels PA, Borst P. Telomere conversion in trypanosomes. Nucleic Acids Res. 1983 Dec 10;11(23):8149-65. doi: 10.1093/nar/11.23.8149. PMID 6324075
- [Background] Ford TF, Grant DA, Austen BM, Hermon-Taylor J. Intramucosal activation of pepsinogens in the pathogenesis of acute gastric erosions and their prevention by the potent semisynthetic amphipathic inhibitor pepstatinyl-glycyl-lysyl-lysine. Clin Chim Acta. 1985 Jan 15;145(1):37-47. doi: 10.1016/0009-8981(85)90017-8. PMID 3919969